CLINICAL TRIAL: NCT02962492
Title: An Investigation Into the Effect of Dapagliflozin on Ketogenesis in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Paresh Dandona, SUNY Distinguished Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1973
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Evaluate Ketogenic Stress
Keywords: Dapagliflozin; Ketogenesis; Type 1 Diabetes; DKA; ketones; exenatide/Bydureon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Ketosis | interventions — Exenatide; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dapagliflozin Arm: (Active Comparator): dapagliflozin 10mg (oral tablet) and exenatide (5µg acutely)/Exenatide extended release (long term) placebo (subcutaneous injection)
  Interventions: Drug: Dapagliflozin
- Exenatide extended release Arm: (Active Comparator): subcutaneous injection of Exenatide (5µg acutely)/Exenatide extended release (long term) and dapagliflozin placebo
  Interventions: Drug: Exenatide/Exenatide extended release
- Placebo Arm: (Placebo Comparator): dapagliflozin placebo (oral tablet) and exenatide (5µg acutely)/Exenatide extended release (long term) placebo (subcutaneous injection)
  Interventions: Drug: Placebo
- Exenatide extended release & dapagliflozin Arm: (Active Comparator): Exenatide (5µg acutely)/Exenatide extended release (long term) and dapagliflozin 10mg
  Interventions: Drug: Exenatide/Exenatide extended release; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Exenatide/Exenatide extended release — Eighty (80) patients with T1D will be enrolled and randomized into 4 groups(20 each) to receive placebo, or dapagliflozin, or exenatide (5µg acutely)/Exenatide extended release (long term), or exenatide (5µg acutely)/Exenatide extended release (long term) and dapagliflozin treatments acutely and for 12 weeks
  Other Names: Bydureon
  Arms: Exenatide extended release & dapagliflozin Arm:; Exenatide extended release Arm:
Drug: Dapagliflozin — Eighty (80) patients with T1D will be enrolled and randomized into 4 groups(20 each) to receive placebo, or dapagliflozin, or exenatide (5µg acutely)/Exenatide extended release (long term), or exenatide (5µg acutely)/Exenatide extended release (long term) and dapagliflozin treatments acutely and for 12 weeks
  Other Names: Farxiga
  Arms: Dapagliflozin Arm:; Exenatide extended release & dapagliflozin Arm:
Drug: Placebo — Eighty (80) patients with T1D will be enrolled and randomized into 4 groups(20 each) to receive placebo, or dapagliflozin, or exenatide (5µg acutely)/Exenatide extended release (long term), or exenatide (5µg acutely)/Exenatide extended release (long term) and dapagliflozin treatments acutely and for 12 weeks
  Other Names: Placebo for both active drugs
  Arms: Placebo Arm:

SUMMARY:
The study investigations include evaluation of the acute effects of a single dose of dapagliflozin (10mg), exenatide (5µg), a combination of exenatide and dapagliflozin or placebo under insulinopenic condition and the long term effect under basal conditions before and after 12 weeks treatment with dapagliflozin, Exenatide extended release, a combination of Exenatide extended release and dapagliflozin or placebo on ketogenesis, glucagon and lipolysis.

DETAILED DESCRIPTION:
The study investigations include evaluation of the acute effects of a single dose of dapagliflozin (10mg), exenatide (5µg), a combination of exenatide and dapagliflozin or placebo under insulinopenic condition and the long term effect under basal conditions before and after 12 weeks treatment with dapagliflozin, Exenatide extended release, a combination of Exenatide extended release and dapagliflozin or placebo on ketogenesis, glucagon and lipolysis.

In the acute effects study, qualified patients will come fasting to the research center. Review of study procedures and vitals will be performed. Insulin infusion (pump) will be stopped and basal blood, urine and adipose tissue biopsy samples will be obtained. Placebos, exenatide (5µg) or dapagliflozin (10mg) (with appropriate placebos) or combination of exenatide and dapagliflozin will be administered, according to a randomized fashion, and blood samples will be collected every 30 min for up to 8 hours after starting the treatment. Urine will be collected every hour up to 8 hours and a second adipose tissue biopsy will be collected at 6 hours after the start of the treatment. Additional blood samples will be collected at 1, 2, 4 and 6 and 8 hour marks for MNC isolation. Plasma and mononuclear cell (MNC) fractions will be prepared from the blood samples. The patient will then come back at the 24 hour mark for a fasting blood and urine collection. The long term study will then commence. Exenatide extended release or dapagliflozin (along with appropriate placebos) or a combination of both drugs will be started and continued for 12 weeks according to original randomization of day 0. In the long term study, dapagliflozin (or the appropriate placebo) will be started at 5mg dose and will be titrated to 10mg/day after 5 days. Fasting blood and 24hr urine samples will be collected at 1, 4 and 8 weeks. At 12 weeks, the 2nd acute effects testing study will be repeated as described above.

Measurements of beta-hydroxybutyrate, acetoacetic acid, glucose, FFA and glucagon, will be measured from all blood samples collected. HSL, GLP-1, glycerol, electrolytes, serum bicarbonate, cortisol and catecholamines will be measured at 0, 60, 120, 240, 360, 480 min and at 24hr following single dose studies at 0 and 12 weeks visits and at baseline on the 1, 4 and 8 weeks visits. Ketone bodies will be measured in all urine samples. All MNC and adipose tissue samples will be tested for HSL and SGLT2 expression.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes for at least 1 year on continuous subcutaneous insulin infusion (CSII; also known as insulin pump)
* HbA1c of 7-10% (inclusive)
* Ages 18-65 years (inclusive of ages 18 and 65)
* BMI 20-30 kg/m2

Exclusion Criteria:

* Inability to give informed consent
* Inability or refusal to comply with protocol
* Use of GLP-1 Receptor Agonists in the last 3 months or DPP-IV and SGLT-2 inhibitors therapy in the last 1 month.
* Risk for pancreatitis (e.g., history of gallstones, alcohol abuse, and hypertriglyceridemia)
* History of pancreatitis and or chronic pancreatitis
* Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) or stroke in the previous 3 months.
* Congestive Heart Failure class III or IV or tachyarrhythmia.
* Hepatic disease: Severe hepatic insufficiency and/or significant abnormal liver function defined as:

  1. Aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
  2. Total bilirubin >2.0 mg/dL (34.2 µmol/L)
  3. Positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody IGM, Hepatitis B surface antigen and Hepatitis C virus antibody
  4. Liver function tests more than 3 times the upper limit of normal
* Renal impairment (e.g., serum creatinine levels ≥1.4 mg/dL for women, or eGFR <60 mL/min/1.73 m2) or history of unstable or rapidly progressing renal disease or end stage renal disease.
* History of unexplained microscopic or gross hematuria, or microscopic hematuria at visit 1, confirmed by a follow-up sample at next scheduled visit.
* HIV positive
* History of gastroparesis
* History of medullary thyroid carcinoma or MEN 2 syndrome
* History of recurring UTI
* Uncontrolled thyroid disease (documented normal TSH), Cushing's syndrome, congenital adrenal hyperplasia or hyperprolactinemia.
* Prior history of a malignant disease requiring chemotherapy or patients with a prior history of bladder cancer regardless of treatment
* Alcoholism or drug addiction.
* Hypertriglyceridemia (>400 mg/dl).
* Any other life-threatening, non-cardiac disease
* Uncontrolled hypertension (BP > 160/95 mm of Hg)
* Patients with hypotension or at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics or recently donated >500ml of blood should have careful monitoring of their volume status
* Pregnant or breastfeeding patients or patient not willing to use two barrier method contraception during study period (unless sterilized or have an IUD)
* Use of hormonal medications, anti-obesity drugs or weight loss medications (prescription or OTC) and medications known to exacerbate glucose tolerance (such as isotretinoin, GnRH agonists, glucocorticoids, anabolic steroids, C-19 progestins) stopped for at least 8 weeks. Use of anti-androgens that act peripherally to reduce hirsutism such as 5-alpha reductase inhibitors (finesteride, spironolactone, flutamide) stopped for at least 4 weeks
* Presence of hypersensitivity to dapagliflozin or other SGLT2 inhibitors (e.g. anaphylaxis, angioedema, exfoliative skin conditions
* Known hypersensitivity or contraindications to use GLP1 receptor agonists (exenatide, liraglutide)
* Known hypersensitivity to heparin/ IV catheter equipment.
* Eating disorders (anorexia, bulimia) or gastrointestinal disorders
* Having a history of bariatric surgery
* Debilitating psychiatric disorder such as psychosis or neurological condition that might confound outcome variables
* Use of an investigational agent or therapeutic regimen within 30 days of study
* Participation in any other concurrent clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes and Endocrinology Research Center of WNY, Williamsville, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin Arm: | Exenatide Extended Release Arm: | Placebo Arm: | Exenatide Extended Release & Dapagliflozin Arm:
Started | 17 | 17 | 13 | 23
Completed | 15 | 15 | 11 | 21
Not Completed | 2 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm: | Dapagliflozin Arm: | Exenatide Extended Release Arm: | Exenatide Extended Release & Dapagliflozin Arm: | Total
Number analyzed (Participants) | 13 | 17 | 17 | 23 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (4.5) | 50.5 (3.2) | 46.5 (3.1) | 44.1 (2.6) | 46.6 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 7 | 11 | 31
  Male | 7 | 10 | 10 | 12 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m²] | 30.8 (1.9) | 28.1 (1.1) | 31.4 (1.8) | 30.7 (1.8) | 30.3 (1.7)
Weight [Mean (Standard Deviation); unit: Kg] | 85.3 (5.8) | 82.6 (3.1) | 91.0 (3.3) | 91.0 (6.0) | 87.9 (5.4)
HbA1c (%) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 7.7 (0.2) | 7.6 (0.2) | 7.5 (0.2) | 7.9 (0.2) | 7.7 (0.2)
daily Basal Insulin Dose/Kg [Mean (Standard Deviation); unit: insulin units/kg] — Basal insulin dose per kg body weight is calculated as number of units of long-acting (basal) insulin treatment needed per day divided by patient weight in kg.
  insulin units/kg | 0.42 (0.08) | 0.40 (0.06) | 0.41 (0.05) | 0.37 (0.03) | 0.40 (0.06)

OUTCOME MEASURES:

1. Primary Outcome: Change in Beta-hydroxybutyrate Levels in Blood
Description: Beta-hydroxybutyrate (BHB) was measured in blood during the acute stress conditions in all the groups after single dose intervention at baseline (0 Week) and at 12 weeks of treatment. The magnitude of change at each of these visits was calculated from each visit baseline (0 hr) and the difference between the change at 12 weeks was compared to the change at 0 week and reported as: Change at week 12 - change at week 0.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: mM
Arm/Group | Placebo Arm: | Dapagliflozin Arm: | Exenatide Extended Release Arm: | Exenatide Extended Release & Dapagliflozin Arm:
Number analyzed (Participants) | 11 | 15 | 15 | 21
mM | -0.23 (0.17) | 0.63 (0.22) | 0.24 (0.21) | 0.31 (0.19)

2. Secondary Outcome: Change in HbA1c Following Treatment
Description: Hemoglobin A1c (HbA1c) was measured in basal conditions in all the groups at week 0 and week 12 of treatment. The change in HbA1c from baseline at 12 weeks is calculated as: HbA1c at week 12 - HbA1c at week 0.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Percent of Hemoglobin (%)
Arm/Group | Dapagliflozin Arm: | Exenatide Extended Release Arm: | Placebo Arm: | Exenatide Extended Release & Dapagliflozin Arm:
Number analyzed (Participants) | 15 | 15 | 11 | 21
Percent of Hemoglobin (%) | -0.3 (0.1) | -0.4 (0.2) | -0.1 (0.1) | -0.9 (0.1)

3. Secondary Outcome: Change in Urinary Beta-hydroxybutyrate (BHB) After 12 Weeks of Treatment
Description: Beta-hydroxybutyrate (BHB) was measured in urine during the acute stress conditions in all the groups after single dose intervention at baseline (0 Week) and at 12 weeks of treatment. The magnitude of change at each of these visits was calculated from each visit baseline (0 hr) and the difference between the change at 12 weeks was compared to the change at 0 week and reported as: Change at week 12 - change at week 0.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: mM
Arm/Group | Placebo Arm: | Dapagliflozin Arm: | Exenatide Extended Release Arm: | Exenatide Extended Release & Dapagliflozin Arm:
Number analyzed (Participants) | 11 | 15 | 15 | 21
mM | 1.2 (0.5) | 0.4 (0.2) | -0.7 (0.6) | 1.1 (0.4)

4. Secondary Outcome: Change in Plasma Glucagon
Description: change in basal plasma glucagon after 12 weeks of dapagliflozin and Bydureon or combination of both treatments compared to baseline
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo Arm: | Dapagliflozin Arm: | Exenatide Extended Release Arm: | Exenatide Extended Release & Dapagliflozin Arm:
Number analyzed (Participants) | 11 | 15 | 15 | 21
pg/ml | 2 (2) | 16 (10) | -15 (8) | -10 (6)

5. Secondary Outcome: Change in Total Insulin Dose
Description: change in total (basal or long acting and short acting) insulin daily dose calculated as daily units/Kg body weight at 12 weeks from baseline (0 week). Long acting or basal insulin dose (in units of insulin) plus short acting (meal) insulin doses administered through the day and reported by patients in patients logs or from insulin pumps are added and divided by body weight in Kg. The reported total insulin dose/Kg represents the average of last 3-7 days before the visit.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Units/Kg
Arm/Group | Placebo Arm: | Dapagliflozin Arm: | Exenatide Extended Release Arm: | Exenatide Extended Release & Dapagliflozin Arm:
Number analyzed (Participants) | 11 | 15 | 15 | 21
Units/Kg | -0.01 (0.02) | -0.02 (0.02) | -0.05 (0.02) | -0.04 (0.02)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Patients were mainly monitored for 2 adverse events (also considered serious adverse events) throughout the study (12 weeks) related to:
  1. severe hypoglycemia (blood sugar <35mg/dl and requiring assistance)
  2. diagnosis of diabetic ketoacidosis
Arm/Group | Placebo Arm: | Dapagliflozin Arm: | Exenatide Extended Release Arm: | Exenatide Extended Release & Dapagliflozin Arm:
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/15 | 0/15 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15 | 0/15 | 0/21
Other Adverse Events (participants affected / at risk) | 0/11 | 0/15 | 0/15 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm: (N=11) | Dapagliflozin Arm: (N=15) | Exenatide Extended Release Arm: (N=15) | Exenatide Extended Release & Dapagliflozin Arm: (N=21)
Severe Hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — severe hypoglycemia (blood sugar <35mg/dl and requiring assistance)
Diabetic Ketoacidosis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Diagnosis or hospitalization due to diabetic ketoacidosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT02962492/Prot_SAP_000.pdf